CLINICAL TRIAL: NCT03146325
Title: Helicobacter Pylori and Body Iron in Adults
Acronym: HEISA
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: Study was not funded and PI has left the institution
Sponsor: The University of Texas Health Science Center, Houston (Other)
Collaborators: Baylor College of Medicine (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: HEISA
Record Dates: First submitted 2017-05-05; First posted 2017-05-09 (Actual); Last update posted 2017-05-09 (Actual); Status verified 2017-05

CONDITIONS: Helicobacter Pylori Infection
Keywords: H. pylori infection

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- PYLERA AND OMEPRAZOLE (Experimental): 14-DAY COURSE OF 3-1 PYLERA (3 CAPSULES QID) PLUS OMEPRAZOLE (BID)
  Interventions: Drug: BISMUTH TETRACYCLINE METRONIDAZOLE OMEPRAZOLE
- PLACEBO (Placebo Comparator): MATCHING PLACEBOS
  Interventions: Drug: MATCHING PLACEBO

INTERVENTIONS:
Drug: BISMUTH TETRACYCLINE METRONIDAZOLE OMEPRAZOLE — A 14-day quadruple Hp eradication therapy consisting of: omeprazole (20 mg twice daily) plus 3 capsules q.i.d., each containing 420 mg of bismuth subcitrate potassium, 375 mg of metronidazole and 375 mg of tetracycline hydrochloride, for 14 days
  Other Names: PYLERA; OTC OMEPRAZOLE
  Arms: PYLERA AND OMEPRAZOLE
Drug: MATCHING PLACEBO — TO BE PREPARED BY LICENSED COMPOUNDING PHARMACY
  Arms: PLACEBO

SUMMARY:
This study is an etiologic trial to test the hypothesis that predicts that Helicobacter pylori eradication in asymptomatic/mildly dyspeptic adults will result in an increase in body iron. The study will assign and aims to complete the follow-up of 240 subjects half of them assigned to a highly effective FDA approved 14-day course of a 3-1 capsule containing bismuth subcitrate, metronidazole and tetracycline plus omeprazole which is now OTC. We have tested the effectiveness of this therapy in the study population and it seems to yield almost 100% eradication on PP analysis. We need the best possible, near 100% eradication rate, which we have already obtained in a pilot, to make comparisons on ITT basis and safely conclude that H pylori leads to a deficit of body iron.

DETAILED DESCRIPTION:
This etiologic double-blind randomized trial in non-anemic mostly asymptomatic/mildly dyspeptic Hp-infected adults will assess whether Hp eradication results in improvements in the levels of iron stores. Iron stores will be assessed by (i) SF as primary outcome, and the following secondary outcomes: (ii) serum transferrin receptor (sTfR), (iii) the ratio of sTfR to SF or R/F, which will be used to estimate body iron, (iv) transferrin saturation (TS), (v) zinc protoporhyrin (ZPP) and (vi) hemoglobin (Hb) at baseline and at 6 months of follow-up. This study is a double-blind randomized clinical trial (RCT) of Hp eradication allocating 400 Hp-infected asymptomatic/mildly dyspeptic adults 18-65 years of age of El Paso, Texas, to receive either (i) a 14-day quadruple Hp eradication therapy described above or (ii) placebo. We expect that at least 240 will complete the study medications and follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Adults 18-65, men and women, residents of the geographic target area in El Paso, Texas, who consent to participate and complete at least 10 days of the study medication.

Exclusion Criteria:

* Unsure if they stay in the area, have a history of allergic reactions to any antibiotic, lack adequate specimen for culture, phenylketonurics, women who are pregnant or unwilling to use 2 modern contraceptive methods during the 2-weeks they take the medications, with a history of heavy menses, anemic, history of peptic ulcer disease or had received Helicobacter eradication therapy or have abnormal lab results for kidney and liver functions tests. Will hold the enrollment for 4 weeks to those taking PPI, bismuth salts and antibiotics, and for 3 months since last blood transfusion or receiving intravenous iron preparations.

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2012-11; Primary Completion 2016-06 (Estimated); Study Completion 2016-08 (Estimated)

PRIMARY OUTCOMES:
Serum Ferritin | 6 months after completing therapy
  Changes from baseline at 6 months after completing therapy, controlled by C-reactive protein

SECONDARY OUTCOMES:
Body Iron | 6 months after completing therapy
  Changes from baseline estimated by the ratio of log base 10 of serum transferrin receptor over serum ferritin
Other markers of iron stores, and erythropoiesis | 6 months after completing therapy
  Changes from baseline transferrin saturation, zinc protoporphyrin to estimate free-erythrocyte protoporphyrin, and hemoglobin

CONTACTS AND LOCATIONS:
Locations (1):
- Sparks Community Center, El Paso, Texas, United States

REFERENCES:
- [Background] Cardenas VM, Prieto-Jimenez CA, Mulla ZD, Rivera JO, Dominguez DC, Graham DY, Ortiz M. Helicobacter pylori eradication and change in markers of iron stores among non-iron-deficient children in El Paso, Texas: an etiologic intervention study. J Pediatr Gastroenterol Nutr. 2011 Mar;52(3):326-32. doi: 10.1097/MPG.0b013e3182054123. PMID 21336159